CLINICAL TRIAL: NCT02194985
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Migalastat Hydrochloride Monotherapy in Subjects With Fabry Disease
Brief Title: Open-Label Extension Study of the Long-Term Effects of Migalastat HCL in Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-042; 2014-002701-38 (EudraCT Number)
Expanded Access: NCT01476163 (Available)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; Galafold; Migalastat; AT1001
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Migalastat HCl 150 mg (Experimental): Migalastat HCl 150 milligram (mg).
  Interventions: Drug: migalastat HCl 150 mg

INTERVENTIONS:
Drug: migalastat HCl 150 mg — Migalastat HCl 150 mg (equivalent to 123 mg migalastat) was provided as capsules in blister packs. One capsule was taken orally every other day.
  Other Names: AT1001; Galafold

SUMMARY:
This is an open-label extension study intended to provide continued treatment with migalastat hydrochloride (HCl) for participants with Fabry disease who completed treatment of a previous migalastat HCl study. The study assessed the long-term safety and effectiveness of migalastat HCl.

ELIGIBILITY:
Inclusion Criteria:

* Participant had completed treatment in a previous study of migalastat HCl given as a monotherapy
* Male and female participant agreed to use protocol-identified acceptable contraception
* Participant was willing to provide written informed consent and authorization for use and disclosure of Personal Health Information (PHI)

Exclusion Criteria:

* Participant's last available estimated glomerular filtration rate (eGFR) in the previous study was <30 milliliter (mL)/minute (min)/1.73 meters squared (m^2); unless there was measured GFR available within 3 months of Baseline Visit, which was >30 mL/min/1.73 m^2
* Participant had undergone, or was scheduled to undergo kidney transplantation or was currently on dialysis
* Participant had a documented transient ischemic attack, stroke, unstable angina, or myocardial infarction within the 3 months before Baseline Visit
* Participant had clinically significant unstable cardiac disease in the opinion of the investigator (for example, cardiac disease requiring active management, such as symptomatic arrhythmia, unstable angina, or New York Heart Association class III or IV congestive heart failure)
* Participant had a history of allergy or sensitivity to AT1001 (including excipients) or other iminosugars (for example, miglustat, miglitol)
* Participant required treatment with Glyset® (miglitol) or Zavesca® (miglustat)
* Participants with severe or unsuitable concomitant medical condition
* Participants with clinically significant abnormal laboratory value(s) and/or clinically significant electrocardiogram (ECG) findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03-14 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Research, Study Director — Amicus Therapeutics
Locations (27):
- United States (7):
  - Clinical Study Site, Atlanta, Georgia
  - Clinical Study Site, Kansas City, Kansas
  - Clinical Study Site, Grand Rapids, Michigan
  - Clinical Study Site, New York, New York
  - Clinical Study Site, Portland, Oregon
  - Clinical Study Site, Dallas, Texas
  - Clinical Study Site, Fairfax, Virginia
- Clinical Study Site, Pilar, Argentina
- Australia (2):
  - Clinical Study Site, Adelaide
  - Clinical Study Site, Parkville
- Clinical Study Site, Vienna, Austria
- Clinical Study Site, Edegem, Belgium
- Clinical Study Site, Porto Alegre, Brazil
- Clinical Study Site, Montreal, Quebec, Canada
- Clinical Study Site, Copenhagen, Denmark
- Clinical Study Site, Cairo, Egypt
- France (2):
  - Clinical Study Site, Garches
  - Clinical Study Site, Lille
- Italy (2):
  - Clinical Study Site, Florence
  - Clinical Study Site, Roma
- Japan (4):
  - Clinical Study Site, Suita, Osaka
  - Clinical Study Site, Niigata
  - Clinical Study Site, Osaka
  - Clinical Study Site, Tokyo
- Clinical Study Site, Barcelona, Spain
- Clinical Study Site, Ankara, Turkey (Türkiye)
- Clinical Study Site, London, United Kingdom

REFERENCES:
- [Derived] Narita I, Ohashi T, Sakai N, Hamazaki T, Skuban N, Castelli JP, Lagast H, Barth JA. Efficacy and safety of migalastat in a Japanese population: a subgroup analysis of the ATTRACT study. Clin Exp Nephrol. 2020 Feb;24(2):157-166. doi: 10.1007/s10157-019-01810-w. Epub 2019 Dec 30. PMID 31889231

RESULTS

PARTICIPANT FLOW:
Groups:
- Migalastat HCl 150 mg: Migalastat hydrochloride (HCl) 150 milligram (mg) was administered orally once every other day for a median duration of 3.1 years (ranged from approximately 1 month to 4.3 years).
Period: Overall Study
Arm/Group | Migalastat HCl 150 mg
Started | 84
Received at Least 1 Dose of Study Drug | 84
Completed | 73
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Met Protocol Defined Stopping Criteria | 3
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All participants who took at least 1 dose of the study drug after they had enrolled into this study.
Groups:
- Migalastat HCl 150 mg: Migalastat HCl 150 mg was administered orally once every other day for a median duration of 3.1 years (ranged from approximately 1 month to 4.3 years).
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 78
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered migalastat that did not necessarily have a causal relationship with the treatment. Each AE was recorded at time of reporting; visits typically occurred every 6 months. Serious AEs were life threatening or resulted in death, resulted in disability/incapacity, hospitalization or prolonged hospitalization, or a congenital anomaly. The criteria for AE severity were: Mild: awareness of sign or symptom, does not interfere with normal everyday activities; Moderate: discomforting, interferes with normal everyday activities, but able to function; Severe: incapacitating, prevents normal everyday activities or significantly affects clinical status and requires medical intervention. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 after first dose to approximately 30 days after last treatment, median duration of 3.1 years
Population: Safety Population: All participants who received at least 1 dose of study drug after they enrolled into this open-label extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 84
Participants
  Participants with at least 1 AE | 80
  Participants with at least 1 serious AE | 26
  Participants discontinued due to AEs | 1
  Participants with AEs leading to death | 0
  Participants with AEs related to study drug | 24
  Participants with AEs unrelated to study drug | 56
  Participants with at least 1 mild AE | 19
  Participants with at least 1 moderate AE | 46
  Participants with at least 1 severe AE | 15

2. Secondary Outcome: Annualized Rate Of Change In The Estimated Glomerular Filtration Rate (eGFR)
Description: The annualized rate of change in the eGFR was assessed per participant by the slope of the simple linear regression between the observed values and the assessment times. It was calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (eGFR [CKD-EPI]) and the Modification of Diet in Renal Disease (MDRD) equation (eGFR [MDRD]). The equations are as follows:
  eGFR [MDRD] = 175 × (1/Serum Creatinine in mg/deciliter^1.154) × (1/Age in years^0.203) × 0.742 [if female] × 1.212 [if black] × 0.808 [if Japanese];
  eGFR [CKD-EPI] = 141 × min(Serum creatinine [Scr]/k, 1)α × max(Scr/k, 1) - 1.209 × 0.993Age × 1.018 [if female] × 1.159 [if black],
  where Scr is serum creatinine, k is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1.
  Participants with at least a Baseline and a post-Baseline value are presented.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: Intent-to-Treat Population: all participants who took at least 1 dose of the study drug after they had enrolled into this study.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 84
mL/min/1.73 m^2
  eGFR[MDRD] | -1.6107 (5.62761)
  eGFR[CKD-EPI] | -1.3528 (4.84795)

3. Secondary Outcome: Change From Baseline In eGFR At End Of Study
Description: The change from baseline in eGFR was calculated using eGFR[CKD-EPI] and eGFR[MDRD] equations. Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of Study was the last recorded observation for each participant (approximately 30 days after last treatment). Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: All participants who took at least 1 dose of the study drug after they had enrolled into this study and had analyzable data at the specified time points.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 82
mL/min/1.73 m^2
  Baseline eGFR[MDRD] | 79.0 (22.56)
  End of Study eGFR[MDRD]: number analyzed (Participants) | 73
  End of Study eGFR[MDRD] | 75.8 (22.90)
  Change from Baseline eGFR[MDRD]: number analyzed (Participants) | 72
  Change from Baseline eGFR[MDRD] | -1.4 (10.62)
  Baseline eGFR[CKD-EPI] | 84.70 (23.092)
  End of Study eGFR[CKD-EPI]: number analyzed (Participants) | 73
  End of Study eGFR[CKD-EPI] | 82.02 (23.890)
  Change from Baseline eGFR[CKD-EPI]: number analyzed (Participants) | 72
  Change from Baseline eGFR[CKD-EPI] | -0.93 (9.828)

4. Secondary Outcome: Change From Baseline In Plasma Globotriaosylsphingosine (Lyso-Gb3) To End Of Study
Description: Concentrations of lyso-Gb3 were measured in plasma using a qualified assay. Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of study was the last recorded observation for each participant (approximately 30 days after last treatment). Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 83
nmol/L
  Baseline | 13.317 (17.5428)
  End of Study: number analyzed (Participants) | 75
  End of Study | 11.758 (16.0662)
  Change from Baseline: number analyzed (Participants) | 75
  Change from Baseline | -1.054 (4.4885)

5. Secondary Outcome: Change From Baseline In White Blood Cell α-Gal A Activity To End Of Study
Description: The activity of the α-galactosidase A (α-Gal A) enzyme was measured in leukocyte lysate by a validated fluorometric assay method, using 4-methylumbelliferone as a reference. The activity values obtained were normalized to protein (measured using a colorimetric assay). Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of Study was the last recorded observation for each participant (approximately 30 days after last treatment). Results for male participants are reported. Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: All male participants who took at least 1 dose of the study drug after they had enrolled into this study and had analyzable data at the specified time points.
Measure: Mean (Standard Deviation); unit: nmol/hr/mg
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 30
nmol/hr/mg
  Baseline: number analyzed (Participants) | 27
  Baseline | 6.882 (6.6857)
  End of Study | 5.290 (5.4054)
  Change from Baseline: number analyzed (Participants) | 24
  Change from Baseline | -1.375 (3.3432)

6. Secondary Outcome: Change From Baseline In 24-hour Urine Protein To End Of Study
Description: A 24-hour urine sample was collected to measure 24-hour urine protein. Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of Study was the last recorded observation for each participant (approximately 30 days after last treatment). Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 83
mg/day
  Baseline | 478.9 (948.59)
  End of Study: number analyzed (Participants) | 66
  End of Study | 394.0 (547.77)
  Change from Baseline: number analyzed (Participants) | 66
  Change from Baseline | 5.4 (233.49)

7. Secondary Outcome: Change From Baseline In Left Ventricular Mass (LVM) To End Of Study
Description: LVM was measured by echocardiography. Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of Study was the last recorded observation for each participant (approximately 30 days after last treatment). Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 70
gram
  Baseline | 178.879 (78.6761)
  End of Study: number analyzed (Participants) | 25
  End of Study | 157.896 (47.9947)
  Change from Baseline: number analyzed (Participants) | 24
  Change from Baseline | -0.803 (18.8522)

8. Secondary Outcome: Change From Baseline In Left Ventricular Mass Index (LVMi) To End Of Study
Description: LVMi was measured by echocardiography. Baseline was defined as the data collected at Month 0, if not available, it was the last visit of the previous (feeder) study if done within 6 months. End of Study was the last recorded observation for each participant (approximately 30 days after last treatment). Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 84
g/m^2
  Baseline: number analyzed (Participants) | 68
  Baseline | 96.513 (36.5691)
  End of Study: number analyzed (Participants) | 25
  End of Study | 83.912 (22.7633)
  Change from Baseline | -0.809 (11.8056)

9. Secondary Outcome: Change From Baseline In Patient Reported Quality Of Life To End Of Study, As Assessed By The Short Form-36 (SF-36) Questionnaire
Description: The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health). Scores on each item are summed and averaged (range: 0=worst to 100=best). Scores were normed to the US population. Higher score indicates less disability. A positive change from baseline indicates improvement. Baseline was defined as the data collected in the last visit of the previous (feeder) study. Only participants with both a Baseline value and an End of Study value were included in the change from baseline analysis.
Time Frame: Baseline to approximately 30 days after last treatment, median duration of 3.1 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 84
units on a scale
  Baseline Physical Functioning | 48.313 (9.2345)
  End of Study Physical Functioning: number analyzed (Participants) | 75
  End of Study Physical Functioning | 46.415 (10.2466)
  Change from Baseline Physical Functioning: number analyzed (Participants) | 75
  Change from Baseline Physical Functioning | -1.276 (7.1627)
  Baseline Role Physical | 46.197 (10.0761)
  End of Study Role Physical: number analyzed (Participants) | 75
  End of Study Role Physical | 45.929 (10.5723)
  Change from Baseline Role Physical: number analyzed (Participants) | 75
  Change from Baseline Role Physical | 0.390 (7.3500)
  Baseline Bodily Pain | 46.889 (10.5983)
  End of Study Bodily Pain: number analyzed (Participants) | 75
  End of Study Bodily Pain | 46.737 (10.3368)
  Change from Baseline Bodily Pain: number analyzed (Participants) | 75
  Change from Baseline Bodily Pain | 0.425 (8.1342)
  Baseline General Health | 44.016 (10.2497)
  End of Study General Health: number analyzed (Participants) | 75
  End of Study General Health | 42.352 (10.1185)
  Change from Baseline General Health: number analyzed (Participants) | 75
  Change from Baseline General Health | -0.811 (5.8672)
  Baseline Vitality | 46.375 (11.8451)
  End of Study Vitality: number analyzed (Participants) | 75
  End of Study Vitality | 45.429 (12.4340)
  Change from Baseline Vitality: number analyzed (Participants) | 75
  Change from Baseline Vitality | -0.674 (8.5076)
  Baseline Social Functioning | 47.433 (10.4985)
  End of Study Social Functioning: number analyzed (Participants) | 75
  End of Study Social Functioning | 47.648 (9.5165)
  Change from Baseline Social Functioning: number analyzed (Participants) | 75
  Change from Baseline Social Functioning | 0.401 (8.4356)
  Baseline Role Emotional | 47.547 (10.3897)
  End of Study Role Emotional: number analyzed (Participants) | 75
  End of Study Role Emotional | 46.141 (10.9054)
  Change from Baseline Role Emotional: number analyzed (Participants) | 75
  Change from Baseline Role Emotional | -0.929 (10.6679)
  Baseline Mental Health | 48.501 (10.6878)
  End of Study Mental Health: number analyzed (Participants) | 75
  End of Study Mental Health | 49.578 (10.5732)
  Change from Baseline Mental Health: number analyzed (Participants) | 75
  Change from Baseline Mental Health | 0.872 (6.2528)
  Baseline Physical Component | 46.184 (10.2268)
  End of Study Physical Component: number analyzed (Participants) | 75
  End of Study Physical Component | 44.825 (10.4292)
  Change from Baseline Physical Component: number analyzed (Participants) | 75
  Change from Baseline Physical Component | -0.508 (6.2494)
  Baseline Mental Component | 47.917 (11.5480)
  End of Study Mental Component: number analyzed (Participants) | 75
  End of Study Mental Component | 48.175 (10.9497)
  Change from Baseline Mental Component: number analyzed (Participants) | 75
  Change from Baseline Mental Component | 0.187 (8.2714)

ADVERSE EVENTS:
Time Frame: Baseline to up to 4.4 years (includes safety follow-up)
Groups:
- Migalastat HCl 150 mg: Migalastat HCl 150 mg was administered orally every other day.
Arm/Group | Migalastat HCl 150 mg
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 26/84
Other Adverse Events (participants affected / at risk) | 74/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat HCl 150 mg (N=84)
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Device malfunction (General disorders) | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Heart rate increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Lipomatosis (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Air embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat HCl 150 mg (N=84)
Palpitations (Cardiac disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 7
Vertigo (Ear and labyrinth disorders) | 7
Hypothyroidism (Endocrine disorders) | 5
Nausea (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 16
Oedema peripheral (General disorders) | 12
Pyrexia (General disorders) | 9
Pain (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 17
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 12
Influenza (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 9
Bronchitis (Infections and infestations) | 6
Overdose (Injury, poisoning and procedural complications) | 12
Albumin urine present (Investigations) | 6
Blood uric acid increased (Investigations) | 6
Protein urine present (Investigations) | 6
Blood creatinine increased (Investigations) | 5
Glomerular filtration rate decreased (Investigations) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Tendonitis (Musculoskeletal and connective tissue disorders) | 7
Paraesthesia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 10
Migraine (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 5
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 6
Proteinuria (Renal and urinary disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Hypotension (Vascular disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02194985/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02194985/SAP_001.pdf